CLINICAL TRIAL: NCT01944176
Title: The Effects of Simvastatin on Th17 Cytokines and Th17 Polarizing Cytokines in COPD Patients
Brief Title: The Effects of Simvastatin on Th17 Cytokines and Th17 Polarizing Cytokine in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Kittipong Maneechotesuwan, Professor, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si323/2013
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: COPD
Keywords: COPD; Statins; Cytokines
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Simvastatin; ubenimex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): simvastatin 20 mg/d is randomized to treat COPD patients for 4 weeks
  Interventions: Drug: simvastatin, placebo
- B1-6-12 (Placebo Comparator): B1-6-12 one tablet a day is randomized to give to COPD patients for 4 weeks
  Interventions: Drug: simvastatin, placebo

INTERVENTIONS:
Drug: simvastatin, placebo
  Other Names: Bestatin; B1-6-12

SUMMARY:
Airway inflammation is partly driven by Th17 and Th17-polarizing cytokines that is steroid-resistant. Statins could suppress IL-17 cytokines in other diseases such as atherosclerosis and multiple sclerosis in mouse model. The investigators hypothesize that statins might provide anti-inflammatory benefit of suppressing IL-17 cytokines in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD without an exacerbation within 3 months prior to study entry
* mild, moderate and severe COPD with or without treatments, regardless of COPD medications

Exclusion Criteria:

* Concomitant other chronic lung diseases including with TB and malignancy
* HIV
* Being on immunosuppressive drugs and systemic corticosteroids
* Dyslipidemic patients with recent cardiovascular or cerebrovascular disease within 6 month prior to study entry
* Cognitive impairment
* Currently on macrolides, azole anti-fungal agents, amiodarone and amlodipine

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sputum cytokines | Up to 4 weeks

SECONDARY OUTCOMES:
FEV1 | Up to 4 weeks
Sputum neutrophils | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kittipong Maneechotesuwan, MD., PhD., Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, BKK, Thailand

REFERENCES:
- [Derived] Maneechotesuwan K, Wongkajornsilp A, Adcock IM, Barnes PJ. Simvastatin Suppresses Airway IL-17 and Upregulates IL-10 in Patients With Stable COPD. Chest. 2015 Nov;148(5):1164-76. doi: 10.1378/chest.14-3138. PMID 26043025